CLINICAL TRIAL: NCT01255852
Title: Phase 4 of Atorvastatin for Preventing Occlusion and Restenosis After Intracranial Artery Stenting
Brief Title: Atorvastatin for Preventing Occlusion and Restenosis After Intracranial Artery Stenting
Acronym: APORIAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Xinfeng Liu, Atorvastatin for Preventing Occlusion and Restenosis After Intracranial Artery Stenting, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JLH2
Record Dates: First submitted 2010-12-03; First posted 2010-12-08 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: CVD
Keywords: atorvastatin; intracranial artery stenting; restenosis
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin group (Experimental): Patients in atorvastatin group will received 40 mg atorvastatin daily from 3 days before the index procedure to 12 months after the procedure.
  Interventions: Drug: atorvastatin
- Control group (No Intervention): Patients in control group will receive 20mg atorvastatin daily treatment.

INTERVENTIONS:
Drug: atorvastatin — Patients in atorvastatin group will received 80 mg atorvastatin daily from 3 days before the index procedure to 12 months after the procedure.
  Arms: Atorvastatin group

SUMMARY:
Severe intracranial atherosclerosis with concomitant stenosis is responsible for approximately 10% of all strokes. Retrospective studies have indicated that up to 50% of patients with a recently symptomatic intracranial stenosis experience recurrent ischemic events. Due to the high stroke risk, patients with high grade 70% symptomatic intracranial stenosis represent the main target group for endovascular treatment. Atorvastatin is widely used in the treatment of hyperlipidemia, especially after acute myocardial infarction. High-dose atorvastatin has been known to stop the progression of atherosclerosis and to decrease the levels of inflammatory markers. Several recent clinical trials have proved atorvastatin can reduce restenosis after stent implantation in coronary artery. But the feasibility of atorvastatin in preventing restenosis in patients with intracranial stenting has not been evaluated.The purpose of this prospective, randomized, single-blinded trial is to evaluate the effect of atorvastatin 80 mg daily in preventing restenosis and related vascular events in patients with intracranial stent implantation.

DETAILED DESCRIPTION:
Severe intracranial atherosclerosis with concomitant stenosis is responsible for approximately 10% of all strokes. In Asian populations intracranial stenoses are even the most commonly found vascular lesions. Retrospective studies indicated that up to 50% patients with recently symptomatic intracranial stenosis experienced recurrent ischemic events. The risk of recurrent stroke increases with the aggravation of intracranial artery stenosis. In Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) trial, 14% and 23% of the patients with TIA or stroke attributable to high-grade intracranial stenosis had further ipsilateral ischemic stroke over the next year despite best medical treatments. If percentage of intracranial stenosis exceeded 70%, the stroke risk went up to 20% in the first year. These results spurred the enthusiasm for endovascular approaches, including percutaneous transluminal balloon angioplasty (PTA) and stenting to treat this potentially harmful disease. Due to the high stroke risk, patients with high-grade ≥70% symptomatic intracranial stenosis represent the main target group for endovascular treatment.

Endovascular management of intracranial arthrosclerosis is, however, associated with an appreciable number of potential complications, including local thrombosis, thromboembolism and, especially, restenosis and in-stent occlusion. To date, the reported 1-year restenosis rates after intracranial stenting in case series and small trials have varied widely, ranging from less than 10% in some to more than 50% in others. According to a recent review, the overall 1-year restenosis rate of intracranial stenting was 25%, and the in-stent occlusion rate was nearly 10%. These relatively high rates of restenosis and re-occlusion after procedure have raised the question about whether stenting improves the natural course of intracranial atherosclerosis.

Compared with the relatively good durability of angioplasty and stenting procedures within the extracranial carotid artery, the high incidence of restenoses appears to be a major drawback of intracranial stenting. Recent studies suggested that especially younger patients treated with self-expandable stents within the anterior circulation have a higher risk for this complication. Considering about 33% of restenoses were symptomatic (TIA or stroke), decreasing restenosis rates after intracranial stenting became the key issue for improving the clinical feasibility of this treatment strategy.

Animal studies have indicated that statins can inhibit platelet aggregation and release of platelet-derived mediators, reduce inflammatory responses of vascular wall, improve artery endothelial function, all of which may contribute to decrease proliferative responses after stent implantation. These profiles make statin optimal for preventing restenosis or occlusion after intracranial stenting, but this strategy has not been tested by clinical trials to date, although statin has been proved by several recent clinical trials to be efficacious in preventing restenosis after stent implantation in coronary arteries.

The initial attempts to lower restenosis rates after coronary balloon angioplasty have failed to demonstrate beneficial effects of statin therapy, although the FLuvastatin Angioplasty REstenosis (FLARE) trial reported a reduction in mortality and myocardial infarction in the fluvastatin treatment patients. Subsequent studies, however, did confirm that statin therapy can decrease restenosis rates and the related ischemic events after stent implantation in patients with coronary artery diseases. Unlike chronic vessel shrinkage may account for ≥70% of recurrence rates after balloon angioplasty, restenosis after coronary stent implantation is entirely due to neointimal proliferation. Experimental studies have shown that statins are capable of inhibiting intimal proliferation after arterial injury. Results from other studies suggested that statins interfere with proliferative responses after coronary stent implantation in humans. Statin therapy was associated not only with a significant reduction in late lumen loss, but also with a greater net gain after coronary stent implantation. Thus, the discrepancy of the effects of statin therapy on restenosis development after balloon angioplasty compared with coronary stent implantation may be easily reconciled by the different mechanisms underlying the recurrence of luminal narrowing.

Elevated LDL cholesterol levels increase platelet and red-cell aggregability, and thrombosis is believed to have a decisive role in the process of restenosis and in-stent occlusion. Lowering LDL cholesterol levels decreases rates of restenosis in the rat-carotid model, whereas treatment with statin decreases the progression of disease in the rabbit-iliac model independently of an effect on LDL cholesterol. In contrast, in the overstretched-swine-coronary model, no relation between either LDL cholesterol or statin and restenosis was observed. An attempt was made to resolve these conflicts with a prospective clinical study in which 157 patients were treated with or without statin. The results indicated that the rate of restenosis was 12 percent with and 44 percent without statin. More than one study also identified the diagnosis of hypercholesterolemia at the time of coronary stent implantation as a major independent predictor for reduced recurrence rates. But a recent study indicated that statin therapy was associated with a comparable reduction of restenosis rates in patients with average serum cholesterol levels at baseline, suggest that the observed effects are not only due to reduced serum cholesterol levels, but also may be related to the non-lipid anti-atherosclerotic properties of statins.

Since the efficacy of high dose statin in preventing restenosis after coronary artery stenting has been confirmed by several clinical trials, it is reasonable to presume that high-dose statin is also efficacious in preventing restenosis and in-stent occlusion after intracranial stenting, because these two vasculatures share very similar anatomical profiles. The present study is aimed to evaluate the preventive effects of atorvastatin 80 mg daily in decreasing restenosis in a consecutive series of patients undergoing intracranial stent implantation at a single center. The hypotheses of this study is that patients with atorvastatin therapy is associated with improved clinical outcome and reduced restenosis rates 12 months after intracranial stent implantation than patients without atorvastatin therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1: Clinical inclusion criteria

  1. Subject is ≥18 years old
  2. Eligible for percutaneous endovascular intervention
  3. Documented severe (70%) symptomatic intracranial stenosis
  4. Acceptable candidate for intracranial stenting
  5. Subject (or legal guardian) understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
  6. Subject willing to comply with all specified follow-up evaluations
* 2: Angiographic Inclusion Criteria

  1. Target lesion located in intracranial internal artery, intracranial vertebral artery, basilar artery or middle cerebral artery
  2. Target lesion must be symptomatic
  3. Target lesion diameter stenosis ≥70%
  4. Reference vessel diameter (RVD): ≥2.0 mm to ≤6.0 mm
  5. Cumulative target lesion length (area to be treated must be completely coverable by one study stent) ≤30 mm
  6. Target lesion is presumed accessible by endovascular treatment.
  7. One non target lesion may be treated in a non target vessel
  8. Non-target lesion in non-target vessel must be treated with a commercially available stent.
  9. Treatment of a non target lesion (if performed) must be deemed a clinical angiographic success, without requiring use of unplanned additional stent(s).
  10. Treatment must be completed prior to treatment of target lesion

Exclusion Criteria:

* Contraindication to ASA, or to both clopidogrel and ticlopidine
* Known hypersensitivity to atorvastatin
* Known allergy to stainless steel
* Known allergy to platinum
* Previous treatment of the target vessel with angioplasty
* Previous treatment of the target vessel with stent
* Previous treatment of any non target vessel with stent within 9 months of the index procedure
* Planned endovascular treatment to post index procedure
* Planned or actual target vessel treatment with an unapproved device, directional or rotational intracranial atherectomy, laser, cutting balloon or transluminal extraction catheter immediately prior to stent placement
* Cerebral infarction within 1 month prior to the index procedure
* Myocardial infarction within the past 1 month
* Uncontrollable malignant hypertension (>180/110 mmHg) before procedure
* Acute or chronic renal dysfunction (creatinine > 2.0 mg/dl or 177 μmol/l)
* Anticipated treatment with atorvastatin or other statins during the 12 months after the index procedure
* Any prior true anaphylactic reaction to contrast agents; defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure
* Leukopenia (leukocyte count < 3.5 × 109/liter)
* Thrombocytopenia (platelet count < 100,000/mm3)
* Thrombocytosis (> 750,000/mm3)
* Seizure 12 months before procedure
* Intracranial tumor
* Active peptic ulcer or active gastrointestinal (GI) bleeding
* Male or female with known intention to procreate within 12 months after the index procedure
* Positive pregnancy test within 7 days before the index procedure, or lactating
* Life expectancy of less than 24 months due to other medical conditions
* Co-morbid condition(s) that could limit the subject's ability to comply with study follow-up requirements or impact the scientific integrity of the study
* Currently participating in another investigational drug or device study
* Current treatment, or past treatment within 6 months with atorvastatin or other statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | at two year
  Target lesion failure (TLF) will be conducted in-hospital and planned at 30 days, 3 months, 6 months, and 12 months. In-stent late diameter loss and stent patency will be evaluated by DSA (digital subtraction angiography) 12 months after the index procedure.

SECONDARY OUTCOMES:
Clinical endpoint | at two years
  Clinical endpoint measurements, TIA, minor stroke, ipsilateral stroke, major stroke, myocardial infarction, cardiovascular death and death, will be conducted in-hospital and planned at 30 days, 3 months, 6 months, and 12 months.
Angiographic follow-up | at two years
  Angiographic follow-up is planned at 3 and 9 months after the index procedure with TCD or CTA for evaluating in-stent blood flow velocity and stent patency.
In-segment binary restenosis rate 12 months after the index procedure | at two years
  In-segment binary restenosis rate 12 months after the index procedure will be evaluated with DSA.
Effects of atorvastatin on blood lipid and inflammatory levels | at two years
  Effects of atorvastatin on blood lipid and inflammatory levels will be evaluated by testing serum CRP, LDL, HDL and MMP-9 at baseline and at 12 month after the index procedure.
Effects of atorvastatin treatment on neurological function outcomes | at two years
  Effects of atorvastatin treatment on neurological function outcomes will be evaluated by mRS,NIHSS,MMSE (modified Rankin Scale,an scale used to assess levels of neurological impairment; The National Institute of Health stroke scale, a standardized method used by physicians and other health care professionals to measure the level of impairment caused by a stroke; mini-mental state examination, a brief 30-point questionnaire test that is used to screen for cognitive impairment) tested 1, 3, 6, 9 and 12 months after the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, MD, Study Chair — Department of Neurology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Department of Neurology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China